CLINICAL TRIAL: NCT06051227
Title: Fentanyl or Esketamine for Traumatic PAIN (FORE-PAIN) Trial
Acronym: FORE-PAIN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Stichting ZiektekostenVerzekering Krijgsmacht (Unknown); Ambulance Amsterdam (Unknown)
Responsible Party: Principal Investigator, Robert Weenink, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP-2023; 2022-500176-63-00 (Other: EU Clinical Trials Information System); U1111-1287-7486 (Other: ICTRP); 2022-000039-22 (EudraCT Number)
Record Dates: First submitted 2023-09-13; First posted 2023-09-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain Due to Trauma; Analgesia; Fentanyl; Esketamine; Emergency Medical Services
Keywords: Analgesics; Ketanest; Administration, intranasal; Administration, intravenous; Pain management; Drug-Related Side Effects and Adverse Reactions; Anesthetics
MeSH Terms: conditions — Agnosia; Drug-Related Side Effects and Adverse Reactions | interventions — Fentanyl; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fentanyl IV (Active Comparator): Opioid analgesic Form: fentanyl solution for injection/infusion Administration: intravenous Initial dose: 1 ug/kg Second dose (if required): 0.6ug/kg
  Interventions: Drug: Fentanyl Citrate
- Fentanyl IN (Experimental): Opioid analgesic Form: fentanyl solution for injection/infusion Administration: intranasal using nasal atomizer Initial dose: 1.25 ug/kg to a maximum of 100ug Second dose (if required): 1ug/kg to a maximum total dose of 2ug/kg
  Interventions: Drug: Fentanyl Citrate
- Esketamine IV (Experimental): Anesthetic, in lower doses the analgesic effect is dominant Form: esketamine solution for injection/infusion Administration: intravenous Initial dose: 0.2mg/kg Second dose (if required): 0.12mg/kg
  Interventions: Drug: Esketamine
- Esketamine IN (Experimental): Anesthetic, in lower doses the analgesic effect is dominant Form: esketamine solution for injection/infusion Administration: intranasal using a nasal atomizer Initial dose: 0.625mg/kg to a maximum of 50mg Second dose (if required): 0.5mg/kg to a maximum total dose of 1mg/kg
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Fentanyl Citrate — Subjects receive one dose of study medication (fentanyl or esketamine) at baseline, either intravenous or intranasal
  Arms: Fentanyl IN; Fentanyl IV
Drug: Esketamine — Subjects receive one dose of study medication (fentanyl or esketamine) at baseline, either intravenous or intranasal
  Arms: Esketamine IN; Esketamine IV

SUMMARY:
Fentanyl and esketamine are both standard of care for treatment of acute severe traumatic pain in the prehospital setting in the Netherlands. However, it is not known whether they are equally effective and safe. It is also not known whether intranasal (IN) administration of fentanyl or esketamine is equally effective and safe as intravenous (IV) administration.

The FORE-PAIN trial is a double-blind multi-arm randomized non-inferiority trial comparing Fentanyl IN, esketamine IV and esketamine IN (intervention arms) to fentanyl IV (comparator arm) for prehospital management of traumatic pain. The investigators hypothesize that all intervention arms provide analgesia that is non-inferior to the comparator arm, and that all study arms are equally safe.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* pain has been caused by a trauma (any trauma mechanism) that occurred on the same day
* Emergency Medical Services personnel determines that administration of a strong opioid or esketamine for analgesia is required
* patient will be transported to a hospital

Exclusion Criteria:

* (estimated) weight <40 or >100 kg
* subject does not understand Dutch or English
* inability to report pain score
* inability to give IN or IV medication
* known severe cardiovascular disease
* pre-eclampsia
* Glasgow Coma Scale score < 11
* subject is known to have previously declined participation in medical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in pain score as measured with Numeric Rating Scale (NRS) | 10 minutes after first drug administration
  NRS is an 11 point Likert scale ranging from 0 to 10, where 0 means 'no pain' and 10 means 'worst pain imaginable'

SECONDARY OUTCOMES:
Change in pain score as measured with NRS | 20 minutes after first drug administration; time of arrival at the hospital (expected within 30 minutes after first drug administration)
  NRS is an 11 point Likert scale ranging from 0 to 10, where 0 means 'no pain' and 10 means 'worst pain imaginable'
Relative change in pain score as measured with NRS | 10 and 20 minutes after first drug administration; time of arrival at the hospital (expected within 30 minutes after first drug administration)
  NRS is an 11 point Likert scale ranging from 0 to 10, where 0 means 'no pain' and 10 means 'worst pain imaginable'
Number of subjects requiring a second dose of study medication | 10 and 20 minutes after first drug administration
  If the patient requires additional analgesia, study medication can be repeated once
Patient satisfaction with pre-hospital analgesia | Time of arrival at the hospital (expected within 30 minutes after first drug administration)
  Patient satisfaction is measured using an 11 point Likert scale ranging from 0 to 10, where 0 means 'extremely unsatisfactory' and 10 means 'extremely satisfactory'
Number of patients experiencing adverse events | Up to time of arrival at the hospital (expected within 30 minutes after first drug administration)
  Including side effects
Number of patients requiring unblinding | Up to time of arrival at the hospital (expected within 30 minutes after first drug administration)
  E.g. because of treatment failure or side effects

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Prof. dr. dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Ambulance Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Metadata and final data will be published. Conditions for reuse apply.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Metadata are published before locking of the database. The final data are published at the time of the journal article's publication.
Access Criteria: Conditions for reuse of data are described in the patient information folder. Access to the data can be granted by the Principal Investigator based on these criteria.

REFERENCES:
- [Derived] de Grunt MN, Risvanoglu N, Siegers JA, Kroon MAGM, Merkus MP, Hollmann MW, Ridderikhof ML, Weenink RP. Fentanyl or esketamine for traumatic pain (FORE-PAIN) trial: study protocol for a double-blind multi-arm randomized non-inferiority trial. Trials. 2025 May 26;26(1):172. doi: 10.1186/s13063-025-08869-9. PMID 40420189